CLINICAL TRIAL: NCT04048356
Title: Chlorhexidine Gluconate Versus Povidone Iodine for Vaginal Surgical Preparation for Urogynecological Procedures
Brief Title: Chlorhexidine vs. Iodine for Vaginal Preparation in Urogynecologic Procedures
Acronym: CLNUP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-039
Record Dates: First submitted 2019-08-02; First posted 2019-08-07 (Actual); Results first posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Pelvic Organ Prolapse; Urinary Incontinence; Pelvic Floor Disorders; Gynecologic Disease; Post-Op Infection; Surgical Site Infection; Urinary Tract Infections
Keywords: Urogynecology; Surgery; Antiseptic Preparation
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence; Pelvic Floor Disorders; Genital Diseases, Female; Surgical Wound Infection; Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be anesthetized during the intervention and will not be informed of the arm of their randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chlorhexidine gluconate (Experimental): Chlorhexidine gluconate 2% vaginal scrub, to be applied vaginally and perineally immediately prior to surgery.
  Interventions: Drug: Vaginal scrub, to be applied vaginally and perineally immediately prior to surgery.
- Povidone Iodine (Active Comparator): Povidone iodine vaginal scrub, to be applied vaginally and perineally immediately prior to surgery.
  Interventions: Drug: Vaginal scrub, to be applied vaginally and perineally immediately prior to surgery.

INTERVENTIONS:
Drug: Vaginal scrub, to be applied vaginally and perineally immediately prior to surgery. — Vaginal scrub, to be applied vaginally and perineally immediately prior to surgery.

SUMMARY:
This is a randomized controlled trial to determine if there is a difference between chlorhexidine gluconate and povidone iodine vaginal preparations for urogynecological surgery post operative infections.

DETAILED DESCRIPTION:
The purpose of this randomized controlled trial is to determine whether there is a difference in efficacy of two of the most common commercially available vaginal surgical preparations. The first objective is to determine whether chlorhexidine gluconate is non-inferior to povidone iodine with respect to post-operative infections including urinary tract infections (both culture proven and empirically treated) and surgical site infections (as defined by the Centers for Disease Control). The second objective is to determine whether chlorhexidine gluconate is non-inferior to povidone iodine with respect to vulvar and vaginal irritation.

ELIGIBILITY:
Inclusion Criteria:

* Female Subjects >18 years of age
* English or Spanish speaking/reading
* Must be able to provide informed consent
* Undergoing urogynecologic procedures or surgery

Exclusion Criteria:

* Pregnant - all patients are verified regarding pregnancy status prior to gynecologic surgical intervention at all sites of surgery - for patients who are premenopausal and have a uterus, a urine pregnancy test is administered in the preoperative setting. Pregnancy status is also determined prior to this in the office setting by interview and patient provided history prior to offering surgery to the patient.
* Inability to return for follow-up visits
* No concurrent need for vaginal antisepsis, such as cases of sacral neuromodulation
* Lack of telephone
* Known allergy to either antiseptic agent
* Prisoners will not be eligible to participate in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Taylor, BA, Study Director — University of New Mexico
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rockefeller NF, Petersen TR, Komesu YM, Meriwether K, Dunivan G, Ninivaggio C, Jeppson PC. Chlorhexidine gluconate vs povidone-iodine vaginal antisepsis for urogynecologic surgery: a randomized controlled noninferiority trial. Am J Obstet Gynecol. 2022 Jul;227(1):66.e1-66.e9. doi: 10.1016/j.ajog.2021.12.260. Epub 2021 Dec 29. PMID 34973179

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chlorhexidine Gluconate | Povidone Iodine
Started | 72 | 65
Completed | 61 | 58
Not Completed | 11 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chlorhexidine Gluconate | Povidone Iodine | Total
Number analyzed (Participants) | 61 | 58 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (13) | 57 (12) | 57.5 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 58 | 119
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 0 | 2 | 2
  White | 30 | 20 | 50
  Latinx | 26 | 25 | 51
  American Indian | 5 | 12 | 17
  Other | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 61 | 58 | 119

OUTCOME MEASURES:

1. Primary Outcome: Rate of Urinary Tract Infection
Description: Urinary tract infection as defined by positive urine culture of >10,000 cfu, or empirically treated symptoms.
Time Frame: 2 weeks post operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine Gluconate | Povidone Iodine
Number analyzed (Participants) | 61 | 58
Participants | 4 | 7

2. Secondary Outcome: Rate of Surgical Site Infection
Description: Surgical site infection as defined by CDC guidelines: https://www.cdc.gov/nhsn/pdfs/pscmanual/9pscssicurrent.pdf
Time Frame: 14 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine Gluconate | Povidone Iodine
Number analyzed (Participants) | 61 | 58
Participants | 1 | 2

3. Secondary Outcome: Vaginal Irritation
Description: Vaginal irritation (including specific symptoms of discomfort, burning, or itching) based on a 5-point scale (Likert type, from 0 minimum/better to 5 maximum/worse, total score reported))
Time Frame: Post operative day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine Gluconate | Povidone Iodine
Number analyzed (Participants) | 54 | 54
Participants
  Vaginal irritation - 0 | 50 | 50
  Vaginal irritation - 1 | 1 | 0
  Vaginal irritation - 2 | 1 | 0
  Vaginal irritation - 3 | 0 | 2
  Vaginal irritation - 4 or 5 | 2 | 2

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Chlorhexidine Gluconate | Povidone Iodine
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/58
Serious Adverse Events (participants affected / at risk) | 4/61 | 4/58
Other Adverse Events (participants affected / at risk) | 0/61 | 0/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chlorhexidine Gluconate (N=61) | Povidone Iodine (N=58)
Surgical Site Infection (Infections and infestations) | 1 (1) | 2 (2)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Bronchitis
Suture reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — suture abscess
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — self-limited delayed vulvar skin irritation 72 hours after surgery
Bacterial Vaginosis (Infections and infestations) | 1 (1) | 0 (0) — BV
Urethral injury (Renal and urinary disorders) | 1 (1) | 0 (0) — urethral injury at the time of aborted midurethral sling placement.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/56/NCT04048356/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/56/NCT04048356/ICF_001.pdf